CLINICAL TRIAL: NCT01641926
Title: A Multicenter Open-label Study to Evaluate the Safety and Efficacy of PEG-Intron™ Versus PEGASYS™ in Subjects With HBeAg Positive Chronic Hepatitis B and HBeAg Negative Chronic Hepatitis B Protocol No. MK-4031-376-00 (Also Known as SCH 054031, P08450)
Brief Title: A Study of the Safety and Efficacy of Pegylated Inferferon Alfa-2b (PEG-Intron™) Versus Pegylated Interferon Alfa-2a (PEGASYS™) in Participants With Chronic Hepatitis B (P08450)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early due to poor recruitment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08450; MK-4031-376 (Other: Merck study number)
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HBeAg(+) PEG-Intron (Experimental): HBeAg-positive participants receive 1.5 mcg/kg/wk PEG-Intron subcutaneously (SC) once weekly for 48 weeks.
  Interventions: Biological: PEG-Intron™
- HBeAg(+) PEGASYS (Active Comparator): HBeAg-positive participants receive 180 mcg/kg/wk PEGASYS SC once weekly for 48 weeks.
  Interventions: Biological: PEGASYS™
- HBeAg(-) PEG-Intron (Experimental): HBeAg-negative participants receive 1.5 mcg/kg/wk PEG-Intron SC once weekly for 48 weeks.
  Interventions: Biological: PEG-Intron™
- HBeAG(-) PEGASYS (Active Comparator): HBeAg-negative participants receive 180 mcg/kg/wk PEGASYS SC once weekly for 48 weeks.
  Interventions: Biological: PEGASYS™

INTERVENTIONS:
Biological: PEG-Intron™ — PEG-Intron subcutaneously (SC) once weekly for a total of 48 weeks
  Other Names: SCH 054031; Pegylated interferon alfa-2b
  Arms: HBeAg(+) PEG-Intron; HBeAg(-) PEG-Intron
Biological: PEGASYS™ — PEGASYS subcutaneously (SC) once weekly for a total of 48 weeks
  Other Names: Pegylated interferon alfa-2a
  Arms: HBeAG(-) PEGASYS; HBeAg(+) PEGASYS

SUMMARY:
This study is being done to compare the safety and efficacy of PEG-Intron™ to that of PEGASYS™ in participants with chronic hepatitis B (hepatitis B envelope antigen [HBeAg] positive or negative) who have not previously been treated with interferon.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to adhere to dose and visit schedules
* ≥ 40 kg
* Hepatitis B surface antigen (HBsAg) positive for at least 6 months
* Anti-HBs negative
* Female participants of childbearing potential must agree to use an acceptable

method of contraception from at least 2 weeks prior to Day 1 and continue until at least 1 month after last dose of study drug

Inclusion Criteria for HBeAg(+) participants:

* HBeAg(+)
* Anti-HBe(-)

Inclusion Criteria for HBeAg(-) participants:

* HBeAg(-)
* Anti-HBe(+)

Exclusion Criteria:

* Co-infection with the human immunodeficiency virus (HIV) or hepatitis C or hepatitis D virus
* Prior treatment with interferon for hepatitis B
* Use of nucleoside/nucleotide analogues within 6 months of the screening visit or at any time during the study
* Use of any investigational drug within 30 days of the screening visit
* Prior treatment with herbal remedies with known hepatotoxicity. All herbal remedies used for hepatitis B treatment must be discontinued before Day 1
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy
* Diabetic and/or hypertensive with clinically significant ocular examination findings
* History of stroke or transient ischemic attack
* Immunologically mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], celiac disease, rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, sarcoidosis, severe psoriasis requiring oral or injected treatment, or symptomatic thyroid disorder)
* Chronic pulmonary disease (e.g., chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidosis)
* Current or history of any clinically significant cardiac abnormalities/dysfunction
* Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
* Myelodysplastic syndromes
* Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair
* Pregnant or nursing, or intending to become pregnant during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2016-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hepatitis B envelope antigen (HBeAg)-positive or -negative participants who were interferon treatment-naïve were recruited from 81 sites to be randomly assigned to receive pegylated inferferon alfa-2b (PEG-Intron™) or pegylated interferon alfa-2a (PEGASYS™).
Pre-assignment Details: 402 participants were enrolled and 399 participants were treated on study.
Period: Overall Study
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS
Started | 143 | 145 | 57 | 57
Treated (All Participants as Treated) | 142 | 144 | 56 | 57
Completed | 115 | 130 | 46 | 53
Not Completed | 28 | 15 | 11 | 4
Not completed — Adverse Event | 5 | 2 | 3 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0
Not completed — Physician Decision | 6 | 5 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 13 | 5 | 6 | 1
Not completed — Not Treated | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Participants as Treated (APaT: all randomized participants who received ≥1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS | Total
Number analyzed (Participants) | 142 | 144 | 56 | 57 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (7.73) | 33.6 (9.23) | 41.1 (10.77) | 42.0 (10.50) | 35.5 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 43 | 21 | 15 | 133
  Male | 88 | 101 | 35 | 42 | 266
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 142 | 144 | 56 | 57 | 399

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HBeAg(+) Participants Achieving HBeAg Seroconversion at 24 Weeks Post-treatment
Description: Blood samples were drawn to assess the participant's seroconversion status at Follow-up (FU) Week 24. HBeAg seroconversion was defined as loss of HBeAg in HBeAg(+) participants and development of antibody to HBeAg.
Time Frame: FU Week 24 (Study Week 72)
Population: All randomized HBeAg(+) participants who received ≥1 dose of study medication. HBeAg(-) participants were not analyzed for HBeAg seroconversion.
Measure: Number; unit: percentage of participants
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS
Number analyzed (Participants) | 142 | 144 | 0 | 0
percentage of participants | 25.4 | 23.6 |  |
Statistical Analysis 1: Comparison: HBeAg(+) PEG-Intron vs HBeAg(+) PEGASYS; The treatment difference in the rates (PEG-Intron arm minus PEGASYS™ arm) and its 95% confidence interval adjusted for the baseline stratification factor (hepatitis B Virus [HBV] genotype) was computed using the method of Miettinen and Nurminen weighted by stratum sample size; Test type: Superiority or Other; Adjusted Treatment Difference = 1.6, 95% CI 2-sided [-8.4 to 11.6]

2. Primary Outcome: Percentage of HBeAg(-) Participants Achieving Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels <2000 IU/mL at 24 Weeks Post-treatment
Description: The Roche COBAS TaqMan HBV-(High Pure System Assay) was used to measure HBV DNA in blood samples of HBeAg(-) participants. The percentage of HBeAg(-) participants with HBV DNA <2000 IU/mL at 24 weeks post-treatment was reported.
Time Frame: FU Week 24 (Study Week 72)
Population: All randomized HBeAg(-) participants who received ≥1 dose of study medication. HBeAg(+) participants were not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS
Number analyzed (Participants) | 0 | 0 | 56 | 57
percentage of participants |  |  | 30.4 | 33.3
Statistical Analysis 1: Comparison: HBeAg(-) PEG-Intron vs HBeAg(-) PEGASYS; The treatment difference in the rates (PEG-Intron arm minus PEGASYS™ arm) and its 95% confidence interval adjusted for the baseline stratification factor (HBV genotype) was computed using the method of Miettinen and Nurminen weighted by stratum sample size; Test type: Superiority or Other; Adjusted Treatment Difference = -3.0, 95% CI 2-sided [-20.2 to 14.3]

3. Secondary Outcome: Percentage of HBeAg(+) Participants Achieving HBV DNA <2000 IU/mL at 24 Weeks Post-treatment
Description: The Roche COBAS TaqMan HBV-(High Pure System Assay) was used to measure HBV DNA in blood samples of HBeAg(+)participants. The percentage of HBeAg(+) participants with HBV DNA <2000 IU/mL at 24 weeks post-treatment was reported.
Time Frame: FU Week 24 (Study Week 72)
Population: All randomized HBeAg(+) participants who received ≥1 dose of study medication. HBeAg(-) participants were not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS
Number analyzed (Participants) | 142 | 144 | 0 | 0
percentage of participants | 23.9 | 21.5 |  |
Statistical Analysis 1: Comparison: HBeAg(+) PEG-Intron vs HBeAg(+) PEGASYS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted Treatment Difference = 2.6, 95% CI 2-sided [-7.2 to 12.3]

4. Secondary Outcome: Percentage of HBeAg(+) and HBeAg(-) Participants Achieving Alanine Aminotransferase (ALT) Normalization at 24 Weeks Post-treatment
Description: ALT normalization is a desired goal of HBV treatment, which is defined as having abnormal ALT levels at baseline and subsequently normal ALT levels after receiving treatment, where normal is defined as ≤ 1x the upper limit of normal (ULN). The percentage of HBeAg(+) and HBeAg(-) participants achieving ALT normalization at 24 weeks post-treatment was reported.
Time Frame: FU Week 24 (Study Week 72)
Population: All randomized HBeAg(+) and HBeAg(-) participants who received ≥1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS
Number analyzed (Participants) | 142 | 144 | 56 | 57
percentage of participants | 49.3 | 47.2 | 71.4 | 61.4
Statistical Analysis 1: Comparison: HBeAg(+) PEG-Intron vs HBeAg(+) PEGASYS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted Treatment Difference = 2.1, 95% CI 2-sided [-9.5 to 13.6]
Statistical Analysis 2: Comparison: HBeAg(-) PEG-Intron vs HBeAg(-) PEGASYS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted Treatment Difference = 10.1, 95% CI 2-sided [-7.2 to 27.1]

5. Secondary Outcome: Percentage of HBeAg(+) Participants Achieving the Combined Response of HBeAg Seroconversion and HBV DNA <2000 IU/mL at 24 Weeks Post-treatment
Description: HBeAg seroconversion was defined as loss of HBeAg in HBeAg(+) participants and development of antibody to HBeAg. HBV DNA levels in blood were measured by the Roche COBAS TaqMan HBV-(High Pure System Assay). The percentage of HBeAg(+) participants with the combined response of achieving both HBeAg conversion and HBV DNA levels <2000 IU/mL at 24 weeks post-treatment was reported.
Time Frame: FU Week 24 (Study Week 72)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAg(-) PEGASYS
Number analyzed (Participants) | 142 | 144 | 0 | 0
percentage of participants | 14.8 | 13.9 |  |
Statistical Analysis 1: Comparison: HBeAg(+) PEG-Intron vs HBeAg(+) PEGASYS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted Treatment Difference = 0.9, 95% CI 2-sided [-7.4 to 9.2]

ADVERSE EVENTS:
Time Frame: SAEs up to 30 days after Week 24 Post-Treatment Visit (up to 76 weeks) Nonserious AEs up to Treatment Week 48 (up to 48 weeks)
Description: APaT population; all randomized participants who received ≥1 dose of study medication.
Arm/Group | HBeAg(+) PEG-Intron | HBeAg(+) PEGASYS | HBeAg(-) PEG-Intron | HBeAG(-) PEGASYS
Serious Adverse Events (participants affected / at risk) | 12/142 | 10/144 | 1/56 | 2/57
Other Adverse Events (participants affected / at risk) | 126/142 | 124/144 | 50/56 | 50/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBeAg(+) PEG-Intron (N=142) | HBeAg(+) PEGASYS (N=144) | HBeAg(-) PEG-Intron (N=56) | HBeAG(-) PEGASYS (N=57)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBeAg(+) PEG-Intron (N=142) | HBeAg(+) PEGASYS (N=144) | HBeAg(-) PEG-Intron (N=56) | HBeAG(-) PEGASYS (N=57)
Neutropenia (Blood and lymphatic system disorders) | 12 (18) | 13 (17) | 5 (9) | 2 (3)
Vision blurred (Eye disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 11 (19) | 8 (19) | 4 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 12 (15) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 5 (7) | 4 (5) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6) | 9 (15) | 1 (1) | 3 (3)
Asthenia (General disorders) | 8 (8) | 3 (3) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Fatigue (General disorders) | 37 (38) | 30 (35) | 10 (11) | 9 (12)
Influenza like illness (General disorders) | 17 (84) | 19 (24) | 6 (8) | 11 (13)
Injection site erythema (General disorders) | 11 (11) | 3 (4) | 3 (3) | 2 (2)
Injection site reaction (General disorders) | 9 (9) | 2 (2) | 6 (6) | 0 (0)
Malaise (General disorders) | 2 (2) | 2 (3) | 1 (2) | 5 (10)
Pain (General disorders) | 9 (9) | 4 (4) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 66 (116) | 55 (97) | 21 (86) | 20 (35)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (12) | 3 (3) | 2 (4)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5) | 4 (4) | 4 (4)
Alanine aminotransferase increased (Investigations) | 6 (6) | 12 (12) | 1 (1) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (7) | 3 (3) | 3 (3)
Neutrophil count decreased (Investigations) | 6 (16) | 5 (10) | 2 (4) | 4 (11)
Platelet count decreased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 4 (6)
Weight decreased (Investigations) | 9 (10) | 16 (16) | 9 (9) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 17 (19) | 21 (23) | 5 (6) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (20) | 7 (18) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (6) | 3 (6) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 43 (60) | 35 (56) | 21 (29) | 13 (27)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 14 (15) | 13 (24) | 6 (8) | 5 (10)
Headache (Nervous system disorders) | 48 (100) | 35 (94) | 16 (32) | 14 (31)
Depression (Psychiatric disorders) | 8 (8) | 2 (2) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 12 (14) | 10 (16) | 5 (6) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 5 (5) | 6 (7) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (10) | 1 (1) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 57 (57) | 54 (54) | 18 (18) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (13) | 14 (14) | 7 (8) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 12 (12) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts.